CLINICAL TRIAL: NCT05257486
Title: A Post-market Multi-Center Retrospective-Prospective Study to Assess Long-term Clinical Outcomes of Non-melanoma Skin Cancer Patients Treated With eBx
Brief Title: Post-market Multi-Center RETRO-Prospective Study to Assess Long-term Clinical Outcomes NMSC Patients Treated With eBx
Status: Completed | Type: Observational
Sponsor: Xoft, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CTPR-0019
Record Dates: First submitted 2022-02-01; First posted 2022-02-25 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Non-melanoma Skin Cancer
Keywords: NMSC

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- NMSC Treatment: Patients who completed Xoft eBx treatment at least five years from the last treatment.
  Interventions: Device: Xoft eBx

INTERVENTIONS:
Device: Xoft eBx — The Xoft Axxent Electronic Brachytherapy (eBx) System allows for the administration of high dose rate brachytherapy treatments using an electronic source

SUMMARY:
The purpose of this retrospective-prospective study is to evaluate lesions after treatment for BCC or SCC NMSC in order to gain a better understanding of the durability of the treatment, and risk of late toxicities for this patient population.

DETAILED DESCRIPTION:
This is a retrospective-prospective study design. The study is post-market, on-label observational study for the treatment of NMSC. Patients who completed treatment at least five years from the last treatment will be identified and existing data as required by this protocol in the patient's record will be collected in addition to conducting office visits or telehealth visits (video) for long-term follow-up.

The study will include:

Identifying patients, retrospectively, who completed treatment a minimum of five years from the last treatment. The history and demographic data will be collected from up to 300 subjects previously treated with eBx for the treatment of NMSC. Patients will have an office visit or telehealth visit in order for the investigators to assess the lesion site, document absence of recurrence, treatment for recurrence (if applicable), and long-term toxicities at the time of the prospective visit.

ELIGIBILITY:
Inclusion Criteria:

1. Previously completed treatment for non-melanoma skin cancer using Xoft eBx Electronic Brachytherapy System according to standard of care;16
2. Provides informed consent;
3. Greater than 40 years of age;
4. Pathological diagnosis confirmed to be squamous cell carcinoma, or squamous cell carcinoma-in-situ, or basal cell carcinoma prior to treatment;
5. Cancer Staging included in this study:

Stage 0: Tis, N0, M0 Stage 1: T1a, b, c, N0, M0 Stage 2: T2a, N0, M0

Exclusion Criteria:

1. Target area is adjacent to a burn scar;
2. Any prior definitive surgical resection of the cancer, prior to Radiation Treatment;
3. Known perineural invasion;
4. Actinic Keratosis;
5. Known spread to regional lymph nodes;
6. Known metastatic disease;
7. Lesion treated with Mohs surgery.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The first phase of this study will be to identify patients who completed treatment with eBx at least five years ago prior to study onset and collect history and demographic data, and eligibility data retrospectively from the patient records and on source worksheets.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Doggett, MD, Principal Investigator — Mission Health
Locations (2):
- United States (2):
  - Kenneth A. Miller, MD Dermatology, Campbell, California
  - Dermatology & Laser Center of San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: No
No plan not sharing IPD

REFERENCES:
- [Result] Doggett SW, Willoughby M, Miller KA, Mafong E. Long-term clinical outcomes of non-melanoma skin cancer patients treated with electronic brachytherapy. J Contemp Brachytherapy. 2023 Feb;15(1):9-14. doi: 10.5114/jcb.2023.125580. Epub 2023 Feb 28. PMID 36970438
- See also: Long-term clinical outcomes of non-melanoma skin cancer patients treated with electronic brachytherapy — https://doi.org/10.5114/jcb.2023.125580

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NMSC Treatment
Started | 183
Completed | 180
Not Completed | 3
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Population: Subjects with eBx Treatment that completed at least 5 Year Follow-up.
Groups:
- NMSC Treatment: Retrospective review to find subjects post Xoft eBx treatment completed at least 5 years ago to complete 1 long-term prospective visit.
  Xoft eBx: The Xoft Axxent Electronic Brachytherapy (eBx) System allows for the administration of high dose rate brachytherapy treatments using an electronic source
Arm/Group | NMSC Treatment
Number analyzed (Participants) | 180
Age, Continuous [Mean (Standard Deviation); unit: Year] | 82.3 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 176
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 178
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 180

OUTCOME MEASURES:

1. Primary Outcome: Local Recurrence
Description: Physician office visit for long-term assessment to determine if recurrence of skin cancer has occurred at previously treated site for subjects who were previously treated at least 5 years prior; Subjects treated with Xoft eBx or MMS over 5 years prior were called in for a long-term prospective visit, reconsented, and assessed for skin cancer recurrence at the previously treated site.
Time Frame: Retrospective review of subject's post Xoft eBx or MMS treatment completed 5-10 years ago, data assessed during a 1-day long-term prospective clinic visit by study completion.
Population: 180 Patients that completed eBx treatment with at least 5 Year follow-up
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | NMSC Treatment
Number analyzed (Participants) | 180
Number analyzed (Lesions) | 182
Lesions | 2

2. Secondary Outcome: Skin Toxicities
Description: Assessment of treatment site at a long-term follow-up visit conducted at 5 years or greater post treatment to determine if late toxicities have occurred at the previously treated site where either eBx or Mohs was performed. Subjects treated with Xoft eBx or MMS over 5 years prior were called in for a long-term prospective visit, reconsented, and assessed for late toxicities at the previously treated site.
Time Frame: as for outcome 1
Population: Patients who completed Xoft eBx treatment at least five year follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | NMSC Treatment
Number analyzed (Participants) | 180
Participants | 129

ADVERSE EVENTS:
Time Frame: Retrospective review of subject's post Xoft eBx or MMS treatment completed 5-10 years ago, data assessed during a 1-day long-term prospective clinic visit by study completion.
Description: Select Skin toxicity adverse events according to CTCAE.
Arm/Group | NMSC Treatment
All-Cause Mortality (participants affected / at risk) | 0/180
Serious Adverse Events (participants affected / at risk) | 0/180
Other Adverse Events (participants affected / at risk) | 129/180
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NMSC Treatment (N=180)
Hypopigmentation Grade 1 (Skin and subcutaneous tissue disorders) | 120 (120)
Telangiectasia Grade 1 (Skin and subcutaneous tissue disorders) | 41 (41)
Scar Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperpigmentation Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Induration Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT05257486/Prot_SAP_000.pdf